CLINICAL TRIAL: NCT02669667
Title: A Phase 1a Randomized, Blinded, Placebo-controlled, Single-ascending Dose Study to Evaluate the Safety and Tolerability of MEDI9314 in Healthy Adult Subjects
Brief Title: Safety and Tolerability of MEDI9314 as Single Ascending Dose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4361C00002
Record Dates: First submitted 2016-01-20; First posted 2016-02-01 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Safety; Healthy Subjects
Keywords: MEDI9314; Safety; Tolerability; Pharmacokinetics; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): single dose of MEDI9314 or placebo
  Interventions: Drug: MEDI9314; Drug: placebo
- Cohort 2 (Experimental): single dose of MEDI9314 or placebo
  Interventions: Drug: MEDI9314; Drug: placebo
- Cohort 3 (Experimental): single dose of MEDI9314 or placebo
  Interventions: Drug: MEDI9314; Drug: placebo
- Cohort 4 (Experimental): single dose of MEDI9314 or placebo
  Interventions: Drug: MEDI9314; Drug: placebo
- Japanese Cohort (Experimental): single dose of MEDI9314 or placebo
  Interventions: Drug: MEDI9314; Drug: placebo
- Cohort 5 (Experimental): single dose of MEDI9314 or placebo
  Interventions: Drug: MEDI9314; Drug: placebo

INTERVENTIONS:
Drug: MEDI9314 — single dose of MEDI9314
Drug: placebo — single dose of placebo

SUMMARY:
This is a phase 1a randomized, blinded, placebo-controlled, single-ascending dose study to assess the safety and tolerability of MEDI9314 in healthy adult subjects

DETAILED DESCRIPTION:
This is a phase I study to assess the safety, tolerability pharmacokinetics, and immunogenicity of MEDI9314 following single dose administration to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age 18 through 50 years at the time of screening.
3. Female subjects must be of non-childbearing potential.
4. Nonsterilized males who are sexually active with a female partner of childbearing potential must use condom and spermicide.
5. Body mass index of 19.0 through 32.0 kg/m2 at screening.
6. No clinically significant abnormality on the basis of medical/medication history or physical examination.
7. Negative drugs of abuse (DOA).
8. Able and willing to comply with the requirements of the protocol and complete the study until the end of the safety follow up period.
9. For the Japanese Cohort, both of the subject's parents and both sets of grandparents must be Japanese.

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
2. Concurrent enrollment in another clinical study involving any treatment.
3. Individuals who are legally institutionalized.
4. Receipt of > 2 marketed or investigational biologic agents.
5. Receipt of an investigational biologic agent within 4 months or 5 half-lives prior to screening, whichever is longer.
6. Receipt of any investigational non biologic agent within 3 months or 5 half lives prior to screening, whichever is longer.
7. Use of any medication (prescription or over the counter, including herbal remedies) within 14 days or 5 half lives of Day 1, whichever is longer, unless in the opinion of the investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety.
8. Known history of allergy or reaction to any component of the investigational product formulation.
9. History of anaphylaxis following any biologic therapy.
10. Any clinically relevant abnormal findings in physical examination ECG, vital signs, and laboratory parameters.
11. Positive tuberculosis (TB) test (QuantiFERON®-TB Gold In-tube).
12. Positive hepatitis B surface antigen, hepatitis C virus antibody or HIV test at screening.
13. Receipt of live attenuated vaccines 30 days prior to the date of screening.
14. Where donation of blood or blood products was in excess of 500 mL within an 8-week period in the 3 months prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2017-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, FFPM, Principal Investigator — Parexel; Hakop Gevorkyan, MD, Principal Investigator — Parexel
Locations (2):
- Research Site, Glendale, California, United States
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 18Feb2016 to 12Jun2017 in United States and United Kingdom.
Pre-assignment Details: A total of 124 participants were enrolled in the study; of which 80 participants were screen failures. Forty-four participants were randomized to MEDI9314 or placebo" in 7 treatment groups.
Groups:
- Placebo: Participants received a single subcutaneous (SC) or intravenous (IV) (infused using a syringe infusion pump over 60 to 90 minutes) dose of placebo matched to MEDI9314 on Day 1.
- Cohort 1: Participants received a single SC injection of MEDI9314 45 milligram (mg) on Day 1.
- Cohort 2: Participants received a single SC injection of MEDI9314 150 mg on Day 1.
- Cohort 3: Participants received a single SC injection of MEDI9314 300 mg on Day 1.
- Cohort 4: Participants from Japan received a single SC injection of MEDI9314 300 mg on Day 1
- Cohort 5: Participants received a single IV infusion of MEDI9314 300 mg using a syringe infusion pump over 60 to 90 minutes on Day 1. All participants in this group did not receive the complete planned dose as per protocol. The error in operating the infusion pump resulted in receiving a dose of 247.5 mg instead of the intended 300 mg dose.
- Cohort 6: Participants received a single IV infusion of MEDI9314 450 mg using a syringe infusion pump over 60 to 90 minutes on Day 1.
Period: Overall Study
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 12 | 4 | 4 | 6 | 6 | 6 | 6
Completed | 12 | 4 | 4 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The As-treated population included participants who received any study drug and summarized according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (10.2) | 32.0 (12.1) | 28.0 (5.1) | 32.0 (8.6) | 35.0 (5.3) | 31.2 (8.2) | 36.0 (10.5) | 33.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 4 | 4 | 6 | 6 | 6 | 6 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 4 | 4 | 6 | 6 | 5 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 0 | 6 | 1 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 4
  White | 8 | 1 | 4 | 6 | 0 | 4 | 5 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event is any unfavourable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with use of medicinal product, whether or not considered related to medicinal product. Serious adverse event is any AE that resulted in death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug and up to Day 240.
Time Frame: From the start of study drug administration upto Day 240
Population: As-treated population included participants who received any study drug and summarized according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants
  TEAEs | 8 | 4 | 2 | 5 | 4 | 5 | 5
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Electrocardiogram Abnormalities Reported as TEAEs
Description: TEAEs observed in participants with clinically significant ECG abnormalities were reported.
Time Frame: From the start of study drug administration upto Day 240
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities Reported as TEAEs
Description: Vital sign parameters included blood pressure, heart rate, and temperature. TEAEs observed in participants with clinically significant vital signs abnormalities were reported.
Time Frame: From the start of study drug administration upto Day 240
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Physical Examination Abnormalities Reported as TEAEs
Description: Adverse events observed in participants with clinically significant physical abnormalities were assessed.
Time Frame: From the start of study drug administration upto Day 240
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Description: An abnormal laboratory finding which required an action or medical intervention by the investigator, or a finding judged by the investigator as medically significant should be reported as an adverse event. Laboratory evaluation (haematology, serum chemistry and urinalysis) of blood and urine samples were performed.
Time Frame: From the start of study drug administration upto Day 240
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants
  Liver function test increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Transaminases increased | 1 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With TEAEs Related to Injection Site Reactions
Description: Adverse events of special interest observed in participants with clinically significant injection site reaction were assessed.
Time Frame: From the start of study drug administration upto Day 240
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants
  Infusion site bruising | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infusion site erythema | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infusion site pruritus | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Injection site bruising | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Injection site erythema | 2 | 4 | 1 | 5 | 0 | 0 | 0
  Injection site haemorrhage | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Injection site induration | 0 | 0 | 0 | 0 | 4 | 0 | 0
  Injection site pain | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Injection site pruritus | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Injection site warmth | 1 | 0 | 1 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Serum Drug Concentration Versus Time Curves From Zero to Infinity (AUC 0-inf) of MEDI9314
Description: The area under the serum drug concentration versus time curves from zero to infinity of MEDI9314.
Time Frame: Day 1 (predose); at the end of infusion (for IV groups); 24, 48, 72, and 96 hours post dose; and on Days 8, 10, 15, 22, 29, 36, 43, 57, 85, 113, 141, 197, and 240
Population: Pharmacokinetic (PK) population included all participants in the as-treated population who received MEDI9314 and who have detectable post-dosing MEDI9314 serum concentrations for accurate estimation of PK parameters. The "Number Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: µg*d/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6
µg*d/mL | 3.01 (NA) — Only 2 out of 4 participants had sufficient elimination data for calculating those PK parameter in Cohort 1. Standard deviation of the mean was not provided when having <=2 parameter values. | 68.8 (47.3) | 179 (105) | 264 (159) | 668 (132) | 1440 (126)

8. Secondary Outcome: Area Under the Serum Drug Concentration Versus Time Curve, to Last Quantifiable Time Point (AUClast)
Description: The area under the serum drug concentration versus time curve, to last quantifiable time point of MEDI9314.
Time Frame: as for outcome 7
Population: The PK population included all participants in the as-treated population who received MEDI9314 and who have detectable post-dosing MEDI9314 serum concentrations for accurate estimation of PK parameters. The "Number Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg*d/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6
μg*d/mL | 2.94 (NA) — Only 2 out of 4 participants had sufficient elimination data for calculating those PK parameter in Cohort 1. Standard deviation of the mean was not provided when having <=2 parameter values. | 68.6 (47.3) | 178 (105) | 264 (159) | 667 (132) | 1439 (126)

9. Secondary Outcome: Maximum Observed Serum Drug Concentration (Cmax) of MEDI9314
Description: The maximum observed serum drug concentration of MEDI9314.
Time Frame: as for outcome 7
Population: PK population included all participants in the as-treated population who received MEDI9314 and who have detectable post-dosing MEDI9314 serum concentrations for accurate estimation of PK parameters.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6
µg/mL | 0.425 (0.367) | 5.44 (2.77) | 10.4 (5.63) | 14.1 (8.87) | 79.0 (14.8) | 108 (9.99)

10. Secondary Outcome: Time to Maximum Observed Serum Drug Concentration (Tmax) of MEDI9314
Description: The time to maximum observed serum drug concentration of MEDI9314.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Median (Full Range); unit: Day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6
Day | 4.00 [3.99 to 4.00] | 8.07 [2.99 to 9.03] | 5.52 [3.00 to 9.13] | 5.51 [3.99 to 9.08] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04]

11. Secondary Outcome: Terminal Phase Elimination Half-life (t1/2) of MEDI9314
Description: Terminal phase elimination half-life of MEDI9314
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6
Day | 1.74 (NA) — Only 2 out of 4 participants had sufficient elimination data for calculating those PK parameter in Cohort 1. Standard deviation of the mean was not provided when having <=2 parameter values. | 3.55 (0.685) | 4.72 (0.998) | 5.03 (1.13) | 7.31 (1.29) | 8.95 (1.14)

12. Secondary Outcome: Serum Concentrations of MEDI9314
Description: Baseline indicates the last assessment prior to first dose. For this study, the lower limit of quantification (LLOQ) for MEDI9314 serum concentrations were 19.53 μg/mL. Where serum concentrations were below this value, a serum concentration of 9.770 μg/mL was imputed.
Time Frame: Baseline (Day 1 [predose]) and Day 240
Population: PK population included all participants in the as-treated population who received MEDI9314 and who have detectable post-dosing MEDI9314 serum concentrations for accurate estimation of PK parameters. The "Number Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6
μg/mL
  Baseline | 21.495 (14.790) | 9.770 (0.000) | 22.577 (31.370) | 9.770 (0.000) | 9.770 (0.000) | 9.770 (0.000)
  Day 240: number analyzed (Participants) | 4 | 4 | 6 | 6 | 5 | 6
  Day 240 | 23.432 (20.738) | 9.770 (0.000) | 9.770 (0.000) | 13.167 (8.320) | 9.770 (0.000) | 14.573 (11.766)

13. Secondary Outcome: Number of Participants Positive for Anti-Drug Antibodies to MEDI9314
Description: Blood samples for immunogenicity assessment included the determination of anti-drug antibodies (ADA) for MEDI9314. The number of participants with positive serum antibodies to MEDI9314 were presented.
Time Frame: Baseline (Day 1 [predose]) and Day 240
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 6 | 6
Participants
  Baseline ADA positive | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 240- ADA positive: number analyzed (Participants) | 12 | 4 | 4 | 6 | 6 | 5 | 6
  Day 240- ADA positive | 0 | 0 | 0 | 2 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: From the start of study drug administration upto Day 240
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 8/12 | 4/4 | 2/4 | 5/6 | 4/6 | 5/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6) | Cohort 6 (N=6)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 4 (4) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 3 (5)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.